CLINICAL TRIAL: NCT06927882
Title: Effects of Whole Body Vibration Therapy on Cognitive Function, Balance, and Quality of Life in Older Adults With Mild Cognitive Impairment: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effects of Whole Body Vibration Therapy on Cognitive Function, Balance, and Quality of Life in Older Adults With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Fahad Alanazi, Assistant professor, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JoufU1
Record Dates: First submitted 2025-04-06; First posted 2025-04-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Impairment; Balance; Quality of Life
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WBV Therapy Group (Experimental): * Frequency: 3 sessions per week for 12 weeks.
  * Duration: 25 minutes per session.
  * Vibration Parameters: Participants will undergo whole body vibration therapy at a frequency of 30 Hz, for 25 minutes per session, 3 times a week, with an amplitude of 1-2 mm, over a duration of 12 weeks.
  Interventions: Other: WBV Therapy Group; Other: Control
- Placebo Group (Placebo Comparator): • Participants will stand on a non-vibrating platform and perform similar static and dynamic exercises for the same duration. The platform will mimic the active intervention's noise and display settings to maintain blinding.
  Interventions: Other: Placebo Group:
- Control Group (No Intervention): Only assessment at baseline, after 12 weeks and 6 months.

INTERVENTIONS:
Other: WBV Therapy Group — * Frequency: 3 sessions per week for 12 weeks.
  * Duration: 25 minutes per session.
  * Vibration Parameters: Participants will undergo whole body vibration therapy at a frequency of 30 Hz, for 25 minutes per session, 3 times a week, with an amplitude of 1-2 mm, over a duration of 12 weeks.
  Arms: WBV Therapy Group
Other: Placebo Group: — • Participants will stand on a non-vibrating platform and perform similar static and dynamic exercises for the same duration. The platform will mimic the active intervention's noise and display settings to maintain blinding.
  Arms: Placebo Group
Other: Control — Only assessment at baseline, after 12 weeks and 6 months.
  Arms: WBV Therapy Group

SUMMARY:
This is a double-blind, randomized controlled trial comparing WBV therapy with a placebo intervention and standard care. A total of 150 participants will be recruited and investigated from Prince Mutib Hospital. Participants will be randomly allocated to one of three groups: WBV therapy, placebo (non-vibrating platform), or control (standard care). The study duration will be 12 weeks, with assessments conducted at baseline, post-intervention (12 weeks), and at a 6-month follow-up.

Protocol Parameters Summary

* Session Frequency: 3 times per week.
* Session Duration: 25 minutes per session.
* Vibration Frequency: 30 Hz.
* Amplitude: 1-2 mm.
* Program Duration: 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years and older.
* Diagnosed with mild cognitive impairment (Montreal Cognitive Assessment (MoCA) score of 18-25). One point is added if years of education are less than 12 years[2].
* Able to stand independently or with minimal assistance.
* No contraindications for WBV therapy or exercise.

Exclusion Criteria:

* Diagnosis of dementia.
* Severe musculoskeletal or neurological disorders.
* Implanted electronic medical devices (e.g., pacemaker).
* Inability to comprehend study instructions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) for Cognitive Function | 6 months
  Assessed using the standard Arabic version of the Montreal Cognitive Assessment (MoCA) at baseline, 12 weeks, and 6 months. The tool is a reliable and valid instrument to detect MCI among the elderly. The maximum score is 0-30, with higher scores indicating better cognitive functioning. A score below 26 typically suggests cognitive impairment. These tests evaluate changes in executive function, attention, and overall cognitive ability. The investigator will use the standard Arabic version used among community dwelling Saudi Arabians population with changes in some word to make it suitable for the Arabic speaking Saudi Arabian population

SECONDARY OUTCOMES:
Berg Balance Scale | 6 months
  Balance was assessed using the Berg Balance Scale (BBS), a validated and reliable 14-item tool for measuring functional balance. Each item was scored from 0 to 4, with a maximum total of 56. Higher scores reflect better balance performance. The Arabic-translated version, previously validated for clinical use, was administered at baseline, 12 weeks, and 6 months.
• Quality of Life | 12 weeks
  Health-related quality of life (HRQoL) was measured using the Arabic version of the Short Form-36 Health Survey (SF-36). This self-reported tool comprises 36 items that assess eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Scores for each domain range from 0 to 100, with higher scores indicating better health status. The Arabic version has been culturally adapted and validated for use among Arabic-speaking populations, ensuring both linguistic and conceptual equivalence.
Timed up and go test | 6 month
  Mobility and fall risk were assessed using the Timed Up and Go (TUG) test. Participants were instructed to stand from a seated position, walk 3 meters, turn around, return, and sit down. The time to complete the task was measured in seconds. Higher times indicate reduced mobility and increased fall risk. A TUG time greater than 13.5 seconds is considered indicative of elevated fall risk.

IPD SHARING:
Plan to Share IPD: Undecided